CLINICAL TRIAL: NCT02546700
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Lebrikizumab in Patients With Chronic Obstructive Pulmonary Disease and a History of Exacerbations
Brief Title: A Study to Evaluate Safety and Efficacy of Lebrikizumab in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WB29804; 2015-001122-42 (EudraCT Number)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Lebrikizumab: Biomarker-high (Experimental): Lebrikizumab will be administered subcutaneously once in every 4 weeks up to 24 weeks to the participants considered as biomarker-high.
  Interventions: Drug: Lebrikizumab
- Lebrikizumab: Biomarker-low (Experimental): Lebrikizumab will be administered subcutaneously once in every 4 weeks up to 24 weeks to the participants considered as biomarker-low.
  Interventions: Drug: Lebrikizumab
- Placebo: Biomarker-high (Placebo Comparator): Matching placebo will be administered subcutaneously once in every 4 weeks up to 24 weeks to the participants considered as biomarker-high.
  Interventions: Drug: Placebo
- Placebo: Biomarker-low (Placebo Comparator): Matching placebo will be administered subcutaneously once in every 4 weeks up to 24 weeks to the participants considered as biomarker-low.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab 125 milligrams (mg) will be administered subcutaneously once in every 4 weeks.
  Arms: Lebrikizumab: Biomarker-high; Lebrikizumab: Biomarker-low
Drug: Placebo — Matching placebo will be administered subcutaneously once in every 4 weeks.
  Arms: Placebo: Biomarker-high; Placebo: Biomarker-low

SUMMARY:
Phase II, randomized, double-blind, placebo-controlled, parallel-group clinical trial of lebrikizumab in participants with COPD and a history of exacerbations who are treated with inhaled corticosteroid (ICS) and at least one long-acting bronchodilator inhaler medication. This study will be conducted to assess the safety, efficacy, and patient-reported outcome (PRO) measures.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of COPD greater than or equal to (>/=) 12 months prior to Visit 1
* Post-bronchodilator FEV1/FVC less than (<) 0.70 at Visit 1 or 2
* Post bronchodilator FEV1 <80% predicted at Visit 1 or 2
* Documented history of one or more acute COPD exacerbations requiring treatment with systemic corticosteroids and/or antibiotics or hospitalization within 12 months prior to Visit 1
* Current tobacco smoker or former smoker (having stopped smoking for at least 6 months prior to Visit 1) with a history of smoking >/=10 pack-years (20 cigarettes/day for 10 years)
* On inhaled corticosteroids (ICS) therapy for >/=6 months prior to Visit 1
* On an eligible bronchodilator medication for >/=6 months prior to Visit 1
* Chest X-ray or computed tomography (CT) scan within 6 months prior to Visit 1 or chest X-ray prior to Visit 2 that confirms absence of clinically significant lung disease besides COPD
* Demonstrated adherence with background COPD inhaler medication during screening period
* For female participants of childbearing age, use of single or combined contraceptive methods for the duration of the study

Exclusion Criteria:

* History of severe allergic reaction or anaphylactic reaction to biologic agent or known hypersensitivity to lebrikizumab injection
* History of clinically significant pulmonary disease other than COPD
* Diagnosis of alpha-1-antitrypsin deficiency
* Lung volume reduction surgery or procedure within 12 months prior to Visit 1
* Supplemental oxygen requirement >2 liters/minute (L/min) at rest or with exertion
* Current diagnosis of asthma
* Participants participating in, or scheduled for, an intensive COPD rehabilitation program
* Maintenance oral corticosteroid therapy
* Treatment with systemic corticosteroids within 4 weeks prior to Visit 1 or during screen period
* Unstable ischemic heart disease or other relevant cardiovascular disorders
* Use of an immunomodulatory or immunosuppressive therapy including monoclonal antibodies (includes anti-interleukin-13 (IL) or anti-IL-4/IL-13 therapy)
* Body weight <40 kg
* Any infection that resulted in hospital admission for >/= 24 hours and/or treatment with oral, intravenous (IV), or intramuscular (IM) antibiotics within 4 weeks prior to Visit 1 or during screening
* Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening
* Active parasitic or Listeria monocytogenes infection within 6 months prior to Visit 1 or during screening
* Received a live attenuated vaccine within 4 weeks prior to Visit 1 or during screening
* Active tuberculosis requiring treatment within 12 months prior to Visit 1
* Human immunodeficiency virus (HIV) or other known immunodeficiency
* Hepatitis or known liver cirrhosis
* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ATL), or total bilirubin elevation >/=2.0 x upper limit of normal (ULN) during screening
* Clinically significant abnormality on screening electrocardiogram (ECG) or laboratory tests
* History of alcohol or drug abuse
* Pregnant or lactating

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Absolute Change From Baseline in Pre-bronchodilator Forced Expiratory Volume (FEV1) at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Rate of Moderate or Severe COPD Exacerbation | Baseline up to Week 24
Absolute Change From Baseline in Post-bronchodilator FEV1 at Week 24 | Baseline, Week 24
Absolute Change From Baseline in Pre-bronchodilator FEV1 at Week 24 | Baseline, Week 24
Time to First COPD Exacerbation | Baseline up to Week 24
Change From Baseline in Health-related Quality of Life as Assessed by the Overall Score of the Saint George's Respiratory Questionnaire for COPD (SGRQ-C) at Week 24 | Baseline, Week 24
Change From Baseline in COPD Symptoms as Measured by the Overall Score of the Exacerbations of Chronic Pulmonary Disease Tool (EXACT) at Week 24 | Baseline, Week 24
Change From Baseline in Cough and Sputum as Measured by the Cough and Sputum Domain Score of the EXACT at Week 24 | Baseline, Week 24
Change From Baseline in Dyspnea as Assessed by the Baseline Dyspnea Index/Transition Dyspnea Index (BDI/TDI) at Week 24 | Baseline, Week 24
Percentage of Participants with Adverse Events And Serious Adverse Events | Baseline up to Week 36
Percentage of Participants with Anti-therapeutic Antibody (ATA) to Lebrikizumab | Baseline up to Week 36
Minimum Observed Serum Trough Lebrikizumab Concentration (Cmin) | Pre-dose (Hour 0) at Weeks 4 and 12, at Week 24
Plasma Decay Half-Life (t1/2) | Pre-dose (Hour 0) on Day 1 (Baseline) and Weeks 1, 4, 8, 12, 16, 20; at Weeks 24, 28, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- United States (21):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Phoenix Medical Research Institute, LLC; Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - California Medical Research Associates, Inc., Northridge, California
  - Palmtree Clinical research Inc, Palm Springs, California
  - Finlay Medical Research, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Southeast Regional Res Group, Savannah, Georgia
  - Centex Studies, Lake Charles, Louisiana
  - The Clinical Research Ctr, St Louis, Missouri
  - Comprehensive Clinical Research Inc., Berlin, New Jersey
  - ISA Clinical Research, Jamaica, New York
  - Gastonia Pharmaceutical Research, Gastonia, North Carolina
  - Clinical Research Inst. of Southern Oregon, Pc, Medford, Oregon
  - Piedmont Research Partners LLC, Old Point Station, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - Baylor College of Medicine; Ben Taub Hospital- Guntupalli, Houston, Texas
  - Centex Studies, Houston, Texas
  - Western Washington Medical Group, Everett, Washington
  - Premier Clinical Research, Spokane, Washington
  - MultiCare Health Center of Washington, Tacoma, Washington
- Argentina (5):
  - Centro Médico Dra de Salvo, Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata
  - Centro Respiratorio Quilmes, Quilmes
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Instituto Del Buen Aire, Santa Fe
- Bulgaria (6):
  - Specialized Hospital For Active Treatment of Pneumophthisiatric Diseases; Dept of Pneumonology, Rousse
  - MHC - Sofia, EOOD, Sofia
  - Fifth MHAT - Sofia EAD, Sofia
  - National Multiprofile Transport Hospital Tzar Boris Ill; Clinic of Internal Diseases, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - Medical Center Tara OOD, Veliko Tarnovo
- Canada (4):
  - Concordia Hospital,Repiratory Research, Winnipeg, Manitoba
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Inspiration Research Limited, Toronto, Ontario
- Denmark (3):
  - Hvidovre Hospital, Lungemedicinsk Afdeling, Hvidovre
  - Lungemedicinsk afd. L, Bispebjerg Hospital, København NV
  - Odense Universitetshospital, Lungemedicinsk Forskningsenhed, Odense C
- Hungary (8):
  - Dr. Kenessey Albert Korhaz Es Rendelointezet; Tudoosztaly (Pulmonolgy Dept ), Balassagyarmat
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Selye János Kórház és Rendelőintézet; Allergológiai Szakrendelés, Komárom
  - Matrai Állami Gyógyintézet ; Bronchológia, Mátraháza
  - CRU Hungary Kft, Miskolc
  - Mohacsi Korhaz, Mohács
  - Farmakontroll Bt., Százhalombatta
  - Markusovszky Egyetemi Oktatokorhaz; Tudogondozo, Szombathely
- Mexico (5):
  - Centro de Investigacion y Atencion Integral Durango CIAID, Durango
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Centro Respiratorio de México, México
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro Integral Médico SJR SC, Querétaro
- Poland (5):
  - Mazowieckie Centrum Badan Klinicznych S.C., Grodzisk Mazowiecki
  - Poradnia Pulmonologiczna dla Doroslych, Lódz
  - MS Clinsearch Specjalistyczny NZOZ Janusz Milanowski Katarzyna Szmygin-Milanowska Spółka Jawna, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej PROFILAKTYKA Wladyslaw Pierzchala, Ruda Śląska
  - NZOZ Lekarze Specjalisci, Wroclaw
- Russia (9):
  - FSI Scientific Research Inst, Moscow
  - Central Clinical Hospital #1 of RZhD JCS, Moscow
  - Novosibirsk Municipal Clinical Hospital For Emergency Medicine #2, Novosibirsk
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - LLC Reafan, Novosibirsk
  - LLC Medical Center "Alliance-Biomedical - Russian Group", Saint Petersburg
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - Siberian State Medical University, Tomsk